CLINICAL TRIAL: NCT05237648
Title: Assessing the Effects of Patient Self-Rating of Voice Quality on Voice Therapy Attendance and Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-01409
Record Dates: First submitted 2022-01-21; First posted 2022-02-14 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Dysphonia
MeSH Terms: conditions — Dysphonia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group (Experimental): Participants will complete an online module with content focusing on patient self-rating of vocal quality within 24 hours of evaluation, approximately 1-2 weeks prior to their first therapy session, and within 24 hours after each therapy session;
  Interventions: Other: Online Voice quality education module
- Sham Control Group (Sham Comparator): Participants will complete an online module within 24 hours of evaluation, approximately 1-2 weeks prior to their first therapy session, and within 24 hours after each therapy session with content focusing on vocal hygiene.
  Interventions: Other: Vocal hygiene module
- Control group (No Intervention): Participants will not complete an online module. The groups will be compared in terms of attendance, self-efficacy, and treatment outcome measures based on the data collected within the NYU Voice Center standard of care

INTERVENTIONS:
Other: Online Voice quality education module — The novel online module the authors developed consists of a patient education on acoustic-perceptual rating of voice quality (CAPE-V), practice rating sample recordings of others' voices, and the patient's self-rating of their own voice in real time during a standard sentence-reading task. The module also includes the Self-Efficacy Scale for Voice Therapy.
  Arms: Experimental Group
Other: Vocal hygiene module — The generic online patient education module on vocal hygiene during the waiting period between their initial evaluation and their first therapy session that also includes the Self-Efficacy Scale for Voice Therapy
  Arms: Sham Control Group

SUMMARY:
The purpose of this study is to assess the effects of incorporating educational online modules into voice therapy. One of the main reasons that voice therapy fails is lack of participation and engagement from the patient's side. The researchers hope to learn if increasing patient engagement via educational online modules during this waiting period between evaluation and first therapy session is useful in increasing understanding of the therapeutic framework of voice therapy.

DETAILED DESCRIPTION:
Attendance and adherence are established as consistent challenges in voice therapy. Specific logistical and psychological factors linked to these challenges include the interval between evaluation and initiation of treatment and components of patient motivation. The authors propose a novel online education module involving patient self-ratings of voice quality to be completed at various time points throughout the therapeutic process, including during the waiting period between initial evaluation and first treatment session. The authors hypothesize that completion of this module will increase patient understanding of the conceptual framework of therapy, provide opportunities for inclusion of patient-driven acoustic goals and establish skills in auditory and kinesthetic awareness, which are foundational to behavioral voice therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* English-speaking
* Have access to technology, including Internet
* Diagnosed with dysphonia with a recommended treatment of voice therapy.
* Willingness to complete all clinical/research assessments
* Ability to give informed consent

Exclusion Criteria:

* Patients who undergo surgical intervention during the course of therapy Contraindications for participation in voice therapy
* Diagnosis of Parkinson's Disease or other neurodegenerative, progressive disorder (e.g., ALS)
* Previous training in acoustic-perceptual voice quality rating, for example a speech language pathology student
* Visual impairments that would prevent the completion of an online module.
* Those with self-reported moderate-profound hearing loss or deafness that would preclude them from participating in the study
* Inability to give informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

PRIMARY OUTCOMES:
Change of voice handicap perception across the 3 groups | Baseline (Day 1) visit, 8 - 10 week visit
  Will be measured by Voice Handicap Index -10 (VHI-10), a patient reported outcome measure used to record the patient's perception of impairment or handicap due to a voice problem. A score of over 10 is considered to be abnormal. The scores in all three groups will be compared and analyzed.
Change of Online education module acceptance across the 3 groups | Baseline Visit (Day 1), Last day of visit (up to 4 months from baseline)
  Will be measured by attendance data (number of sessions recommended versus attended, number of no shows) using the standard patient data collected according to standard of care process.

SECONDARY OUTCOMES:
Change of perceived effectiveness of voice therapy | Baseline (Day 1) visit, 8 - 10 week visit
  Self-Efficacy Scale for Voice Therapy will assess a patient's self-perception of their ability to achieve a goal. The Self-Efficacy Scale for Voice Therapy prompts patients to be "brutally honest" and rate their perceived capability to accomplish practice or generalization of skills in various daily and therapeutic situations and activities. Patients are asked to rate their certainty in these capabilities from 0 to 10, where 0 is not at all certain and 10 is extremely certain.
Change of patient's perception on voice therapy | Baseline (Day 1) visit, 8 - 10 week visit
  Comparison of scores on the Patient Perception of Voice Therapy Questionnaire for therapy completers across the three groups as well as between those subjects who completed an online module (experimental and sham control groups) and those who did not (control group alone).
Change of perceptual voice ratings | Baseline (Day 1) visit, 8 - 10 week visit
  CAPE-V will be used to measure experimental group patients and clinician perceptual voice rating. The Consensus Auditory-Perceptual Evaluation of Voice (CAPE-V) indicates salient perceptual vocal attributes, identified by the core consensus group as commonly used and easily understood. The attributes are: (a) Overall Severity; (b) Roughness; (c) Breathiness; (d) Strain; (e) Pitch; and (f) Loudness. The CAPE-V displays each attribute accompanied by a 100- millimeter line forming a visual analog scale (VAS). The clinician indicates the degree of perceived deviance from normal for each parameter on this scale, using a tic mark.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Johnson, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.Upon reasonable request. Requests should be directed to Aaron.Johnson@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.